CLINICAL TRIAL: NCT06953830
Title: Optimal Measurement of Spleen Stiffness Among Veterans With Metabolic Dysfunction-Associated Steatotic Liver Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: William Jennings Bryan Dorn VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nicholas Hoppmann, Physician, William Jennings Bryan Dorn VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1766537-1
Record Dates: First submitted 2025-04-07; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Metabolic-dysfunction-associated Fatty Liver Disease (MAFLD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Spleen Stiffness Measurements (Experimental): Participants with metabolic-dysfunction associated steatotic liver disease will undergo liver and spleen stiffness measurements using vibration-controlled transient elastography
  Interventions: Device: Vibration-controlled transient elastography

INTERVENTIONS:
Device: Vibration-controlled transient elastography — Liver and spleen stiffness measurements using vibration-controlled transient elastography

SUMMARY:
A growing number of people are being diagnosed with fatty liver disease, also known as metabolic-dysfunction associated liver disease (MASLD). Fatty liver disease can unknowingly progress to serious liver disease and even permanent scarring (cirrhosis).The purpose of this research is to learn the best way to detect serious liver disease as early as possible in patients with fatty liver disease by measuring the stiffness of the spleen. Secondarily, the study hopes to understand how the stiffness of the spleen relates to the severity of liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent for participation in a clinical study
* Able to read and comprehend English
* Evidence of fatty liver disease on previous liver biopsy, imaging or clinical documentation

Exclusion Criteria:

* Pregnant
* Known decompensated cirrhosis or hepatocellular carcinoma
* Absence of spleen
* Documentation of alcohol use disorder or alcohol use greater than 20g/day for women or greater than 30 g/day for men
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Spleen Stiffness measurement | 1 year
  Percent of participants with valid spleen stiffness measurements using vibration controlled transient elastography

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hoppmann, MD, Principal Investigator — Columbia VA Healthcare System
Locations (1):
- WJB Dorn VA Medical Center 6439 Garners Ferry Road Columbia, South Carolina 29209, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No